CLINICAL TRIAL: NCT07023432
Title: Belzutifan's Role in Active Surveillance Versus Treatment for Indolentmetastatic Clear Cell Renal Ccell Carcinoma (BRAVE-RCC)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0268; NCI-2025-04261 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-06-10; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Active Surveillance; Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — belzutifan; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Participants will take belzutifan by mouth every day during the study. You will be given a dosing diary to write down when you take each dose of belzutifan, including if you miss or vomit any doses. Bring the diary with you to each visit, along with any leftover study drug and/or study drug bottles.
  Interventions: Drug: Belzutifan
- Observation group (Experimental): Participants will not receive treatment in this study. Instead, you will undergo active surveillance under the discretion of your treating physician.
  Interventions: Other: Active Surveillance

INTERVENTIONS:
Drug: Belzutifan — Given by PO
  Arms: Treatment group
Other: Active Surveillance — Given by Observation
  Arms: Observation group

SUMMARY:
To learn if belzutifan can help to control the disease in patients with metastatic RCC who are considered candidates for active surveillance and have not undergone previous systemic treatment. The safety of belzutifan in this patient population will also be studied.

DETAILED DESCRIPTION:
Primary Objectives

• To compare the progression-free survival difference for participants treated with belzutifan versus active surveillance as evaluated by RECIST 1.1 criteria.

Secondary Objectives

* To describe the safety profile of belzutifan in this population using CTCAE v5.0.
* To estimate the difference in time to start of new systemic treatment in participants treated with belzutifan versus active surveillance.
* To describe objective response rates (CR and PR) using RECIST 1.1 criteria.

Exploratory Objectives

* To describe methylated ctDNA characteristics for participants at baseline, during treatment, and at progression.
* To describe baseline tissue-based gene expression profiling and its association with outcome where tissue is available.
* To estimate differences in target lesion sum of diameters from baseline to start of next systemic therapy.
* To estimate differences in quality of life based on FKSI-19 questionnaire for participants on belzutifan versus surveillance.
* To describe PFS2 (time to second disease progression) in both arms.
* To describe overall survival in both groups.
* To describe the duration of objective response, duration of CR, and duration of SD using RECIST 1.1 criteria.

ELIGIBILITY:
Inclusion Criteria

1. Metastatic clear cell renal cell carcinoma, with or without sarcomatoid features, clinically apparent less than 12 months.
2. Male/female participants must be at least 18 years of age on the day of signing informed consent.
3. IMDC risk score of 0 or 1.
4. No prior systemic treatment for ccRCC. Adjuvant immunotherapy or targeted treatments allowed if progressive disease is noted at least 12 months after last dose of immunotherapy.
5. Metastatic disease that is documented by imaging with CT or MRI and measurable by RECIST1.1.
6. Participants must have signed and dated an Institutional Review Board (IRB)/Institutional Ethics Committee (IEC) approved written informed consent form (ICF) in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal participant care.
7. Karnofsky performance status ≥ 70% and ECOG PS 0 or 1
8. Suitable for active surveillance in the medical judgment of the treating oncologist.
9. Participants must have adequate organ and marrow function as defined below:

   i. absolute neutrophil count ≥ 1.5 x 109/L ii. platelets ≥ 100 x 109/L iii. hemoglobin (Hgb) ≥ 9 g/dL iv. total bilirubin ≤ 1.5 x Institutional upper limit of normal (ULN) v. AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN vi. serum creatinine ≤ 1.5 × institutional ULN OR 24-hour clearance ≥ 40 mL/min

   *Aspartate aminotransferase (serum glutamic-oxaloacetic transaminase)-AST(SCOT)/ Alanine aminotransferase (serum glutamic-pyruvic transaminase)- ALT(SGPT)
10. A minimum of 28 days from any major surgery prior to registration.
11. Ability to swallow, retain, and absorb oral medication.
12. Baseline oxygen saturation >92% on room air.
13. Female Participants are eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

    * Is not a woman of child-bearing potential (WOCBP) OR
    * Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis), during the intervention period and for at least 30 days after the last dose of study intervention. The investigator should evaluate the potential for contraceptive method failure (ie, noncompliance, recently initiated) in relationship to the first dose of study intervention.
    * A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours before the first dose of study intervention.
    * If a urine test cannot be confirmed as negative (eg, an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
    * The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
    * Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
14. Male participants are eligible to participate if they agree to the following during the intervention period and for at least 7 days after the last dose of study intervention:

    * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR
    * Must agree to use contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause as detailed below:

      * Agree to use a male condom plus partner use of an additional contraceptive method when having penile-vaginal intercourse with a WOCBP who is not currently pregnant. Note: Men with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile-vaginal penetration.
      * Male participants must also agree to use male condom when engaging in any activity that allows for passage of ejaculate to another person of any sex.
    * Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
15. Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Exclusion Criteria

1. Known or suspected brain metastases or active leptomeningeal disease.
2. Requires any supplemental oxygen (either intermittent or chronic)
3. Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with protocol
4. Impairment of gastrointestinal function or disease that may significantly alter the absorption of belzutifan (e.g., uncontrolled nausea, vomiting, diarrhea, malabsorption syndromes, prior small bowel resection, or inflammatory bowel disease)
5. Prior cardiovascular event including myocardial infarction, rest claudication, stroke, unstable angina, central nervous system (CNS) hemorrhage, unstable ventricular arrythmias, or severe congestive heart failure (NYHA Class 3 or higher) within the past 6 months
6. Received colony-stimulating factors (eg, granulocyte colony stimulating factor, granulocytemacrophage colony stimulating factor or recombinant erythropoietin) ≤28 days prior to the first dose of study intervention.
7. Has moderate to severe hepatic impairment (Child-Pugh B or C).
8. Participants who have undergone major surgery ≤ 28 days prior to starting study drug, radiation ≤ 2 weeks prior to starting study drug, or who have not recovered from side effects of such therapy prior to registration.
9. Has received any type of small molecule kinase inhibitor (including investigational agents) ≤2 weeks before randomization; any prior HIF-2a antagonist exposure.
10. Has known hypersensitivity or allergy to the active pharmaceutical ingredient or any component of the study intervention (belzutifan) formulations.
11. Is currently receiving either strong (phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate (eg, bosentan, efavirenz, modafinil) inducers of CYP3A4 that cannot be discontinued for the duration of the study.
12. Active infection requiring systemic therapy within 14 days prior to treatment assignment.
13. Has active tuberculosis.
14. Active HBV (defined as HBsAg reactive and detectable HBV viral load) or active HCV (defined as HCV RNA [qualitative] is detected) infection.
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
16. Has uncontrolled HIV infection (history of HIV with CD4 count >400 and undetectable HIV viral load while on anti-retroviral therapy allowed).
17. Pregnant women are excluded from this study. Women who are breastfeeding should discontinue prior to initiating treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-12-03 (Estimated); Primary Completion 2028-04-14 (Estimated); Study Completion 2030-04-14 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org